CLINICAL TRIAL: NCT06693765
Title: A Single Dose, Non-randomised, Open-label, Parallel Group Study to Assess the Pharmacokinetics, Safety, and Tolerability of AZD4144 in Participants With Severe Renal Impairment, End-stage Kidney Disease, and in Healthy Participants
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, and Tolerability of AZD4144 in Participants With Severe Renal Impairment, End-stage Kidney Disease, and in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9440C00003; 2024-513848-28-00 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Renal Impairment; End-stage Kidney Disease; Healthy Participants
Keywords: Intermittent haemodialysis; Chronic kidney disease; Estimated glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1: AZD4144 (Experimental): Participants with severe renal impairment will receive a single oral dose of AZD4144 on Day 1.
  Interventions: Drug: AZD4144
- Cohort 2: AZD4144 (Experimental): Healthy participants with normal renal function will receive a single oral dose of AZD4144 on Day 1.
  Interventions: Drug: AZD4144
- Cohort 3: AZD4144 (Experimental): Participants with ESKD on intermittent haemodialysis will receive a single oral dose of AZD4144 on the first day of Treatment Period 1 and Treatment Period 2.
  Interventions: Drug: AZD4144
- Cohort 4: AZD4144 (Experimental): Participants with moderate renal impairment will receive a single oral dose of AZD4144 on Day 1.
  Interventions: Drug: AZD4144
- Cohort 5: AZD4144 (Experimental): Participants with mild renal impairment will receive a single oral dose of AZD4144 on Day 1.
  Interventions: Drug: AZD4144

INTERVENTIONS:
Drug: AZD4144 — AZD4144 will be administered orally.

SUMMARY:
A study to investigate the pharmacokinetics, safety, and tolerability of AZD4144 in participants with severe renal impairment, end-stage kidney disease, and in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, single dose, non-randomised, parallel group, Phase I study to assess the pharmacokinetics, safety, and tolerability of AZD4144 in male and female participants with severe renal impairment and end-stage kidney disease (ESKD) compared with healthy control participants.

The study will comprise of:

* A Screening Period of 21 days.
* Cohort 1, 2, 4, and 5: a single Treatment Period with an in-clinic period of 7 days.
* Cohort 3: two Treatment Periods each with an in-clinic period of 7 days, and a washout period of 6 days after the in-clinic treatment period.
* A Follow-up visit 7 days following discharge.

ELIGIBILITY:
Inclusion Criteria:

Healthy Matched Control Participants Only (Cohort 2):

* Stable renal function (for example, no clinically significant change in an estimated glomerular filtration rate (eGFR) within 3 months or longer prior to study the Screening Visit), as determined by the investigator.
* Have an eGFR of ≥ 90 milliliter/minute/1.73m2 (mL/min/1.73m2) as determined via the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula without race.

Renally Impaired Participants Only (Cohorts 1, 4 and 5)

* Participants who have renal impairments.
* Cohort 1 participants with severe renal impairment must have an eGFR ≥ 15 to < 30 mL/min/1.73m2 not on dialysis. Cohort 1 should have at least 3 participants with eGFR ≤ 20 mL/min/1.73m2.
* Cohort 4 participants with moderate renal impairment must have an eGFR of ≥ 30 to < 60 mL/min/1.73m2.
* Cohort 5 participants with mild renal impairment must have an eGFR of ≥ 60 to < 90 mL/min/1.73m2.

Cohort 3

* Participants with ESKD on IHD must have been on stable IHD for at least 3 months prior to Visit 1.
* All renally impaired participants should be on stable standard of care for at least 4 weeks prior to Visit 1.

All cohorts:

* Body weight of at least 50 kilograms (kg) and body mass index (BMI) within the range ≥ 18 to ≤ 35 kg/m2, inclusive.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.

Exclusion Criteria:

* History of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* Known history of primary immunodeficiency (congenital or acquired) or an underlying condition that predisposes to infection.
* Concomitant immunosuppressive, steroid treatment.
* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment) (Cohort 2).
* Renal transplant participants, participants on dialysis, and those with a history of acute kidney injury (Cohorts 1, 4, 5).
* Use of any of the prohibited medications in the 4 weeks prior to Visit 1 (Cohorts 1, 3, 4, 5).
* Participants with a known hypersensitivity to AZD4144 or any of the excipients of the product.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUCinf) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Apparent total body clearance (CL/F) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Non-renal clearance of drug from plasma (CLNR/F) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Apparent volume of distribution based on the terminal phase (Vz/F) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Terminal elimination half-life (t½λz) | From Day 1 to Day 14
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Renal clearance of drug from plasma (CLR) | From Day 1 to Day 4
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Amount excreted (Ae) | From Day 1 to Day 4
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.
Percentage of dose excreted unchanged in urine (fe) | From Day 1 to Day 4
  To assess the PK of a single oral dose of AZD4144 in participants with severe renal impairment and ESKD compared with healthy control participants.

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | From Day 1 to Follow-up (Day 14/28)
  To evaluate the safety and tolerability of AZD4144 single dose in participants with severe renal impairment, ESKD, and their healthy controls.

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Sofia, Bulgaria
- Research Site, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. ''Yes", indicates that AZ is accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/